CLINICAL TRIAL: NCT00455325
Title: Genotoxic Stress, Atherosclerosis, and Metabolic Syndrome-AIM 2
Brief Title: Chloroquine to Treat People With Metabolic Syndrome Aim2 (ARCH-MS)
Acronym: ARCH-MS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 395; P50HL083762 (NIH)
Record Dates: First submitted 2007-03-30; First posted 2007-04-03 (Estimated); Results first posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-04

CONDITIONS: Metabolic Syndrome X; Overweight; Hypertension; Dyslipidemias; Prediabetic State
Keywords: Insulin Resistance; Atherosclerosis; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Hypertension; Dyslipidemias; Prediabetic State; Insulin Resistance; Atherosclerosis | interventions — Chloroquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- First Intervention (3 weeks) (Placebo Comparator): Cohort 1: Chloroquine placebo one tablet daily for 3 weeks, followed by 5-7 week rest period.
  Interventions: Drug: Placebo Comparator: First Intervention (3 weeks)
- Second Intervention (3 weeks) (Active Comparator): Cohort 2: 80mg chloroquine or placebo tablet once daily for Weeks 3, followed by 5-7 week rest period.
  Interventions: Drug: Active Comparator: Second Intervention (3 weeks)
- Third Intervention (3 weeks) (Active Comparator): Cohort 3: 80mg chloroquine tablet daily: for 3 weeks, followed by 5-7 week rest period.
  Interventions: Drug: Active Comparator: Third Intervention (3 weeks)
- Fourth Intervention (3 weeks) (Active Comparator): Cohort 4: 250mg chloroquine tablet daily: for 3 weeks, followed by 5-7 week rest period.
  Interventions: Drug: Active Comparator: Fourth Intervention (3 weeks)

INTERVENTIONS:
Drug: Placebo Comparator: First Intervention (3 weeks) — once daily placebo tablet for 3 weeks followed by: euglycemic clamp procedure; 24 hour Ambulatory Blood Pressure; Oral Glucose tolerance Test; serum collection; 24 hour urine collection; collection of peripheral blood mononuclear cells
  Other Names: Placebo once daily
  Arms: First Intervention (3 weeks)
Drug: Active Comparator: Second Intervention (3 weeks) — Once daily 80mg chloroquine or placebo tablet 3 Weeks followed by euglycemic clamp procedure; 24 hour Ambulatory Blood Pressure; Oral Glucose tolerance Test; serum collection; 24 hour urine collection; collection of peripheral blood mononuclear cells
  Other Names: 80 mg chloroquine or placebo tablet once daily
  Arms: Second Intervention (3 weeks)
Drug: Active Comparator: Third Intervention (3 weeks) — Once daily 80mg tablet for 3 weeks followed by: euglycemic clamp procedure; 24 hour Ambulatory Blood Pressure; Oral Glucose tolerance Test; serum collection; 24 hour urine collection; collection of peripheral blood mononuclear cells
  Other Names: 80 mg chloroquine tablet once daily
  Arms: Third Intervention (3 weeks)
Drug: Active Comparator: Fourth Intervention (3 weeks) — Once daily 250mg tablet for 3 weeks followed by: euglycemic clamp procedure; 24 hour Ambulatory Blood Pressure; Oral Glucose tolerance Test; serum collection; 24 hour urine collection; collection of peripheral blood mononuclear cells
  Other Names: 250 mg chloroquine tablet once daily
  Arms: Fourth Intervention (3 weeks)

SUMMARY:
Metabolic syndrome consists of a group of co-occuring conditions that increase an individual's risk of developing heart disease, stroke, and diabetes. The purpose of this study is to evaluate the short-term effectiveness of chloroquine, a protein-activation medication, at improving metabolic syndrome.

DETAILED DESCRIPTION:
Metabolic syndrome is one of the most common disorders in industrialized countries. It consists of abnormal serum lipids, glucose intolerance, elevated blood pressure, and central obesity in the setting of insulin resistance. The syndrome substantially increases the risk of developing diabetes and vascular disease, but there is no clear unifying approach to treat this disorder. In animals, activation of the protein ataxia telangiectasia mutated (ATM) using the antimalarial drug chloroquine improves features of metabolic syndrome and decreases atherosclerosis, a build-up of fatty plaque within arteries. The purpose of this study is to evaluate the effectiveness of short-term treatment with low doses of chloroquine as a way of managing metabolic syndrome.

Participants in this study will initially receive placebo for 3 weeks, followed by increasing doses of chloroquine in three, 3-week intervals. Following each 3-week treatment, participants will be admitted to the research center for one day. There will be a period of no active treatment for 5 to 7 weeks following each admission to the research center to allow recovery from the blood drawing of the clamp procedure before the start of the next treatment interval.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metabolic syndrome, as determined by at least three of the following five criteria:

  1. Elevated fasting triglyceride levels greater than or equal to 150 mg/dL
  2. Low HDL cholesterol levels: less than 50 mg/dL for women and less than 40 mg/dL for men
  3. Hypertension (=>130/85 mm Hg =<160/100 mm Hg) untreated; or hypertension controlled (=<150/90 mm Hg) on a stable medication regimen for 4 weeks prior to baseline visit.
  4. Increased waist circumference: greater than 35 inches in women and greater than 40 inches in men
  5. Elevated fasting glucose levels =<100 mg/dL but =>126 mg/dL
* Subjects may be on a stable doses of a statin drug for at least 3 months
* Subjects may be on a stable doses of L-thyroxine for at least 3 months
* Willing to use acceptable form of birth control (e.g., hormonal birth control, double barrier methods)

Exclusion Criteria:

* Prior travel treatment with chloroquine or hydroxychloroquine as follows:

  1. any exposure in the past 2 years,
  2. >30 days of therapy if exposure was between 2 and 5 years ago,
  3. >90 days of therapy if exposure was between 5 and 10 years ago,
  4. >6 months of therapy if exposure was 10 to 20 years ago,
  5. >1 year of therapy if exposure was 20 to 30 years ago,
  6. No limit if last exposure was >30 years ago, ex. during the Vietnam conflict.
* Morbid obesity (body mass index [BMI] greater than 45)
* Coronary artery disease or other vascular disease
* History of stroke
* Chronic kidney insufficiency (i.e.,estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m2)
* Diabetes
* Seizure disorder
* History of psoriasis
* Blood disorders, including anemia (i.e., hemoglobin levels less than 13 g/dL in men and less than 12 g/dL in women)
* Current malignancy or active treatment for recurrence prevention, example tamoxifen. Cancer considered to be cured, either as a result of surgery or other treatment is not exclusionary.
* Asthma requiring daily beta agonist therapy or intermittent oral steroids is exclusionary. Inhaled steroids are acceptable. Obstructive sleep apnea will be allowed if Continuous Positive Airway Pressure (CPAP) or other therapy has been stable for 6 months. Other active respiratory diseases are excluded.
* Liver disease, or liver function test results greater than twice the normal value
* Active infection, including HIV
* Serious illness requiring ongoing medical care or medication
* Treatment with atypical anti-psychotic medication. Treatment with any other medication for psychiatric illness, unless on a stable dose for 6 weeks prior to enrollment. Patients with unstable psychiatric disorders are excluded per the decision of the study MD regardless of medication history.
* Taking any of the following lipid lowering medications: niacin, fibrates, and greater than 1 gm fish oils
* Uncontrolled hypertension (BP >150/90) at enrollment.
* Need for daily over the counter medications, or currently taking cimetidine or >1000 IU vitamin E daily and unwilling to reduce or discontinue the use of vitamin E or discontinue cimetidine for the duration of the study. Persons taking >1000 IU of vitamin E should reduce the dose 30 days prior to randomization.
* Pregnant, breastfeeding, or intending to become pregnant
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Retinal disease (in particular, drusen or pigmentary changes at the macula); any ocular disease that interferes with the eye examination (e.g., cataracts)
* Auditory disease or hearing loss; persons with total, irreversible hearing loss can be enrolled.
* Participation in another clinical trial within past 30 days prior to screening and 60 days prior to randomization. Questionnaire or observational studies are not exclusionary.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2004-09 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clay F. Semenkovich, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Schneider JG, Finck BN, Ren J, Standley KN, Takagi M, Maclean KH, Bernal-Mizrachi C, Muslin AJ, Kastan MB, Semenkovich CF. ATM-dependent suppression of stress signaling reduces vascular disease in metabolic syndrome. Cell Metab. 2006 Nov;4(5):377-89. doi: 10.1016/j.cmet.2006.10.002. PMID 17084711
- [Derived] McGill JB, Johnson M, Hurst S, Cade WT, Yarasheski KE, Ostlund RE, Schechtman KB, Razani B, Kastan MB, McClain DA, de las Fuentes L, Davila-Roman VG, Ory DS, Wickline SA, Semenkovich CF. Low dose chloroquine decreases insulin resistance in human metabolic syndrome but does not reduce carotid intima-media thickness. Diabetol Metab Syndr. 2019 Jul 29;11:61. doi: 10.1186/s13098-019-0456-4. eCollection 2019. PMID 31384309
- [Derived] Razani B, Feng C, Semenkovich CF. p53 is required for chloroquine-induced atheroprotection but not insulin sensitization. J Lipid Res. 2010 Jul;51(7):1738-46. doi: 10.1194/jlr.M003681. Epub 2010 Mar 5. PMID 20208057
- See also: click here for Washington University Research Participant Registry — https://vfh.wustl.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligibility included adults with at least 3 criteria of metabolic syndrome but who did not have diabetes. Subjects were studied in the setting of a single academic health center. First participant was screened on 08 September 2004. The last study visit occurred on 08 June 2010.
Pre-assignment Details: 144 participants were screened
Groups:
- Placebo Comparator: First Intervention (3 Weeks): Chloroquine placebo one tablet daily for 3 weeks
  Placebo Comparator Limb 1: 1 chloroquine placebo tablet for 3 weeks followed by 5-7 week rest period
- Second Intervention (3 Weeks): 80mg Chloroquine weekly for 3 weeks followed by 5-7 week rest period
- Third Intervention (3 Weeks): 80mg chloroquine tablet daily: for 3 weeks, followed by 5-7 week rest period.
- Fourth Intervention (3 Weeks): 250mg chloroquine tablet daily: for 3 weeks, followed by 5-7 week rest period.
Period: Cohort 1: Placebo
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Started | 35 | 0 | 0 | 0
Completed | 27 | 0 | 0 | 0
Not Completed | 8 | 0 | 0 | 0
Not completed — Started exclusionary drug | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — New diagnosis of Type 2 Diabetes | 1 | 0 | 0 | 0
Not completed — DIFFICULTY WITH IV ACCESS | 1 | 0 | 0 | 0
Period: Cohort 2: 80 mg Chloroquine Weekly
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Started | 0 | 27 | 0 | 0
Completed (This is a sequential study) | 0 | 26 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Period: Cohort 3: 80 mg Chloroquine Daily
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Started | 0 | 0 | 26 | 0
Completed | 0 | 0 | 25 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Started exclusionary drug | 0 | 0 | 1 | 0
Period: Cohort 4: 250mg Chloroquine Daily
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Started | 0 | 0 | 0 | 25
Completed | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized participants, in this sequential, dose escalated study
Groups:
- All Randomized Subject: All Randomized Subjects
Arm/Group | All Randomized Subject
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Full analysis set included all randomized participants
  years | 47 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32
  Black or African American | 3
  Unknown or not reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Hepatic insulin sensitivity was measured by comparing glucose production at baseline of zero insulin infusion rate with glucose production at 56 pmol/m2/min. Hepatic insulin sensitivity was expressed as the percent suppression, such that greater percent suppression indicated greater hepatic insulin sensitivity. There are no reference values, since the patients served as their own controls.
Time Frame: assessed every 8 - 10 weeks at the end of each treatment period
Population: Full Analysis Set included all randomized participants who completed all procedures in the study arm
Measure: Mean (Standard Deviation); unit: % suppression inf rate 56 pmol/m2/min
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
% suppression inf rate 56 pmol/m2/min | .56 (0.04) | 0.55 (0.05) | 0.66 (0.06) | 0.70 (0.04)

2. Secondary Outcome: Systolic Blood Pressure
Description: Two techniques were employed: auscultation of seated subjects at rest was performed by a trained observer who recorded the first and fifth phases of the Korotkoff sounds; and, a portable oscillometric device (SpaceLabs Medical) recorded results every 20 min during the day and every hour during the night. Data were analyzed as mean values over 24 hours.
Time Frame: Assessed every 8-10 weeks at the end of each treatment period
Population: Full Analysis Set included all randomized participants who completed all procedures in the study arm
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mmHg | 121 (12) | 121 (10) | 123 (12) | 123 (12)

3. Secondary Outcome: Diastolic Blood Pressure
Description: as for outcome 2
Time Frame: Assessed every 8-10 weeks at the end of each treatment period.
Population: Full Analysis Set included all randomized participants who completed procedure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mmHg | 70 (7) | 71 (7) | 73 (8) | 73 (9)

4. Secondary Outcome: Total Cholesterol
Description: Fasting Serum Blood Sample
Time Frame: Assessed every 8-10 weeks at the end of each treatment period.
Population: Full analysis set included all randomized participants who completed study procedure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mg/dL | 187 (6) | 181 (7) | 182 (5) | 173 (6)

5. Secondary Outcome: Non-HDL Cholesterol
Description: Fasting Serum Blood Sample
Time Frame: Assessed every 8-10 weeks at the end of each treatment period.
Population: Full Analysis Set included all randomized participants who completed procedure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mg/dL | 144 (6) | 139 (7) | 139 (5) | 131 (6)

6. Secondary Outcome: Low-density Lipoprotein
Description: Fasting Serum Blood Sample
Time Frame: Assessed every 8-10 weeks at the end of each treatment period.
Population: Full Analysis Set included all randomized participants who completed procedure.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mg/dl | 115 (5) | 109 (6) | 109 (5) | 103 (6)

7. Secondary Outcome: Triglycerides
Description: Fasting Serum Blood Sample
Time Frame: Assessed every 8-10 weeks at the end of each treatment period.
Population: Full Analysis Set included all randomized participants who completed procedure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Comparator: First Intervention (3 Weeks) | Second Intervention (3 Weeks) | Third Intervention (3 Weeks) | Fourth Intervention (3 Weeks)
Number analyzed (Participants) | 27 | 26 | 25 | 25
mg/dL | 143 (14) | 153 (16) | 151 (18) | 140 (16)

ADVERSE EVENTS:
Time Frame: From consent date to final visit an average of 4 to 6 months
Description: Safety Analysis Set included all randomized participants
Groups:
- First Intervention: Placebo Comparator (3 weeks) followed by 5-7 week rest period
- Second Intervention: 80mg Chloroquine weekly (3 weeks) followed by 5-7 week rest period
- Third Intervention: 80mg chloroquine daily (3 weeks)followed by 5-7 week rest period
- Fourth Intervention: 250mg chloroquine tablet daily(3 weeks) followed by 5-7 week rest period
Arm/Group | First Intervention | Second Intervention | Third Intervention | Fourth Intervention
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/27 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/27 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 6/35 | 1/27 | 1/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | First Intervention (N=35) | Second Intervention (N=27) | Third Intervention (N=25) | Fourth Intervention (N=25)
IV placement difficulties (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IV infiltration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin reaction to tape (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Extremity erythema due to BP cuff
Vasovagal Syncope (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Vasovagal episode with IV placement
Medication Error (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Incorrect stable isotope administered
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes